CLINICAL TRIAL: NCT06386042
Title: Guideline Implementation and Quality of Care in Patients With Heart Failure: the TITRATE-HF Registry
Acronym: TITRATE-HF
Status: Active, not recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Netherlands Heart Institute (Other)
Responsible Party: Principal Investigator, Jasper Brugts MD PhD, Principal investigator, Dr., Erasmus Medical Center
Other Study IDs: MEC-2022-0252
Record Dates: First submitted 2024-04-17; First posted 2024-04-26 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic heart failure: Patients with chronic HF at least 6 months after the initial HF diagnosis with are in stable condition, treated with HF medication (not necessarily all GDMT) and evaluated for an intrinsic cardiac defibrillator device if applicable.
  Interventions: Other: no intervention, observational study
- Worsening heart failure: Patient with established chronic heart failure which after a period of "stable" HF have experienced an hospital admission with necessity of iv. diuretics or urgent visit needing iv. diuretics. Patients can be included in inpatient / admitted setting or outpatient setting where drug changes during admission (GDMT uptitration) can be recorded. The index event of hospitalisation must be within 6 months prior to inclusion in the registry (retrospective).
  Interventions: Other: no intervention, observational study
- de novo heart failure: Patients with heart failure with reduced ejection fraction (ejection fraction <40% with diagnosis within 3 months of inclusion (de novo heart failure or newly-diagnosed HF) with no previous diagnosis of HF.
  Interventions: Other: no intervention, observational study

INTERVENTIONS:
Other: no intervention, observational study — no intervention, observational registry of the prescription of medical therapy according to the European Society of Cardiology Heart Failure guidelines (quality of care).

SUMMARY:
SUMMARY Rationale: Quality of Care registries provide valuable insight in guideline adherence and implementation of guideline recommendations in routine clinical practice.

Objective: The overall aim of the project is to study the titration of guideline directed medical therapy (GDMT) according to the European Society of Cardiology (ESC) HF 2021 guideline recommendations for patients with heart failure (HF) reduced ejection fraction (HFrEF), and mildly reduced ejection fraction (HFmrEF).

Study design: The current study is a prospective multi-center national quality of care registry (longitudinal) of regular HF care (as given).

Study population: The study population consists of patients with heart failure (de novo HF, chronic HF and worsening HF). Study setting is outpatient or inpatient (during admission). Patient sample is set at a minimum of 4000 patients, but can be expanded during the course of the registry project.

Participating sites: all hospitals with dedicated HF outpatient clinic in the Netherlands can participate.

Data: aggregated data

Intervention: none / no

Main study parameters/endpoints: The main parameters of quality of HF care are the adherence to guideline recommendation in terms of percentage (%) drug prescription, percentage (%) target dose (order, speed) and reason not to adhere to the guideline (intolerance, side-effects, maximum tolerated dose). The main endpoints for prognosis are the number of HF related hospitalizations and all-cause mortality during follow-up.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There is no risk in participation, no intervention and no active involvement of patients for specific activities in the study. The project is a registration of care as given (standard care) to the participating subject with heart failure.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this registry, a subject must meet all of the following criteria:

1. Written informed consent obtained from subject aged ≥18 years.
2. Diagnosis of heart failure according to the European Society of Cardiology 2021 guideline definitions. An eligible patient must also fulfil to the category definitions of de novo HF, chronic HF or worsening HF.
3. Subjects willing and able to comply with the follow-up of regular care at the outpatient clinic. Also, sites should continue regular care for an included subject for at least 1 year (with preferably the entire project) at their outpatient HF clinic in this quality of care project.

Informed Consent: As the current research is a patient file study (registry) without an intervention of any kind. The medical ethics review board has reviewed the study and the study is declared to be not subject to the Medical Research Involving Human Subjects Act. Although informed consent is not strictly necessary, we have decided to ask permission from the patient use to their data for scientific research and comply to privacy/general data protection regulations for scientific research as well as to consent with data-coupling with other official data sources for quality of care projects in the Netherlands.

Exclusion Criteria:

1. Subjects with a life expectancy <1 years due to comorbidities according to the treating physician.
2. Subjects who have had a major cardiovascular event (e.g., myocardial infarction, open heart surgery, stroke) within 2 months interacting with prescription or dosing of HF drugs.
3. Subjects with advanced heart failure (end-stage) scheduled for or likely to undergo heart-transplantation or ventricular assist device within 6 months of baseline visit.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The current registry studies only patient with heart failure and an ejection fraction below 50%.
  Type of heart failure patients
  * Chronic heart failure
  * Worsening heart failure
  * De novo or newly-diagnosed heart failure
Sampling Method: Non-Probability Sample
Enrollment: 4289 (Estimated)
Dates: Start 2022-06-05 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Prescription level (percentage,%) and target dose (percentage, %) of guideline-directed medical therapy for HF | anticipated follow-up is 5 years
  according to European Society of Cardiology guideline recommendations

SECONDARY OUTCOMES:
All-cause mortality | anticipated follow-up is 5 years
  Death
Hospital admission due to heart failure related event and/or urgent visit with necessity of furosemide iv. | anticipated follow-up is 5 years
  Hospitalisation
Hospital admission due to non heart failure related event | anticipated follow-up is 5 years
  Hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf de Boer, Study Chair — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clephas PRD, Malgie J, Schaap J, Koudstaal S, Emans M, Linssen GCM, de Boer GA, van Heerebeek L, Borleffs CJW, Manintveld OC, van Empel V, van Wijk S, van den Heuvel M, da Fonseca C, Damman K, van Ramshorst J, van Kimmenade R, van de Ven ART, Tio RA, van Veghel D, Asselbergs FW, de Boer RA, van der Meer P, Greene SJ, Brunner-La Rocca HP, Brugts JJ. Guideline implementation, drug sequencing, and quality of care in heart failure: design and rationale of TITRATE-HF. ESC Heart Fail. 2024 Feb;11(1):550-559. doi: 10.1002/ehf2.14604. Epub 2023 Dec 8. PMID 38064176